CLINICAL TRIAL: NCT05458778
Title: Detection of Urinary HCG During The Not Pregnancy and Pregnancy Cycles
Brief Title: Detection of Urinary Human Chorionic Gonadotropin (hCG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Quanovate Tech Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022/04/16
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Women who are trying to conceive
  Interventions: Device: Daily test with urine by the product

INTERVENTIONS:
Device: Daily test with urine by the product — Women perform the hCG test and share the test results

SUMMARY:
The Mira Pregnancy Test is an over-the-counter urine hCG test intended for early detection of pregnancy. The test is indicated for use four days before the expected period. Throughout this study, volunteers with non-medical backgrounds were recruited to test hCG with urine samples using the Mira Pregnancy Test during the not pregnancy cycle or pregnancy cycle. To perform the study, a total number of more than 200 volunteers will be recruited to participate in the study.

DETAILED DESCRIPTION:
The studies include two parts, which are a lay user study and a urine samples test during the trying to conceive cycle.

Part 1: Lay user study Part 2: Detection of hCG in Early Pregnancy Clinical Samples

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 and over
* Willing to give informed consent
* Willing to conduct a personal home pregnancy test and reveal their pregnancy status
* Have a working smartphone

Exclusion Criteria:

* Have a medical background or have been in a related industry/occupation
* Volunteers who are unfit to participate in the research by the researcher
* Used the investigational pregnancy test previously
* Has a medical condition
* Confirmed to be pregnant by a healthcare professional and beyond the first trimester (defined as last menstrual period (LMP) +13 weeks)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Include more than 200 worldwide women aged 18 and over taking part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive evaluation via survey and calculating the consistency | From July 2022 to August 2022
  The consistency between the lay-user test results and the actual test results
The accuracy of data was expressed as per the Pregnancy Detection Rate | From July 2022 to August 2022
  The number of positive results on different days obtained by the user of the Mira pregnancy test is divided by the total number of women who confirmed pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MS, Principal Investigator — Quanovate Tech Inc.
Locations (1):
- Quanovate Tech Inc., San Ramon, California, United States